CLINICAL TRIAL: NCT06355778
Title: A Mechanistic Investigation of Risk Factors for Opioid Use Disorder: Examining Hippocampal-based Context-dependent Learning and Memory Associated With Adverse Childhood Experiences
Brief Title: Adversity, Brain and Opioid Use Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Duval, Associate Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00234185; 1R01DA056415 (NIH)
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Healthy
Keywords: Magnetic Resonance Imaging (MRI); Adverse Childhood Experiences; Fear Learning; Memory; Hippocampal function
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opioid use disorder (OUD) group (Other): This group takes buprenorphine and has OUD.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Behavioral: Computer Tasks
- Buprenorphine (BUP) control group: (Other): This group takes BUP and does not have OUD.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Behavioral: Computer Tasks
- Healthy Controls group (Other): This group does not take BUP and does not have OUD.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Behavioral: Computer Tasks

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — Enrolled participants will have one MRI during the study on day 2 after having Day 1 visit. During the MRI the participants will complete various tasks.
Behavioral: Computer Tasks — Eligible participants will complete computer tasks (cognitive tasks, spatial navigation tasks, context dependent fear learning, etc.) at visit 1 and then during the MRI.

SUMMARY:
The way people process and remember information may be related to adverse childhood experiences and Opioid Use Disorder symptoms. The purpose of this project is to examine brain function and performance during learning and memory tasks in adults. The study will compare measures of learning and memory across three groups of participants: those with an Opioid Use Disorder (OUD) that take buprenorphine for opioid replacement therapy, adults without an Opioid Use Disorder taking buprenorphine, and healthy adults that do not have an Opioid Use Disorder and are not taking buprenorphine.

ELIGIBILITY:
Inclusion Criteria for all groups:

* Right handed
* Able to give informed consent
* Normal/corrected-to-normal vision and hearing

Inclusion Criteria for Opioid Use Disorder (OUD) group:

* Diagnosis of OUD
* Be actively receiving buprenorphine (BUP) for opioid agonist therapy
* Be free from illicit substance use for at least 2 weeks
* The study will allow stable dose (> 3 months) of commonly prescribed psychiatric medications and some sleep aids (per protocol)

Inclusion Criteria for the BUP control group:

* Taking BUP for chronic pain
* No Substance Use Disorder (including OUD)
* The study will allow stable dose (> 3 months) of commonly prescribed psychiatric medications and some sleep aids (per protocol)

Inclusion Criteria for Healthy participant group:

* Not taking BUP
* Free of any psychiatric or major medical conditions

Exclusion Criteria for all groups:

* Significant medical or neurologic conditions (e.g., stroke, seizures, multiple sclerosis)
* Actively suicidal
* Contraindication for MRI
* Inability to tolerate small, enclosed spaces without anxiety
* Life history of schizophrenia, bipolar disorder, learning disability, attention deficit disorder, or pervasive developmental disorder
* Use of substances or prescription medications that could interfere with measures of interest (per protocol)
* Unable to provide informed consent
* Participants who have completed other studies in our lab involving learning and memory assessments with the same/similar tasks used here (HUM00230585, HUM00121812) will not be eligible to complete the current study, due to possible learning/practice effects
* Unable to fit comfortably in the MRI scanner due to body size (typically men over 6 feet tall that weigh more than 250 lbs, men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Differences in Blood Oxygen Level Dependent (BOLD) signal in the hippocampus | Day 2 (MRI task visit)
  BOLD signal during functional magnetic resonance imaging (fMRI) will be used as a measure of hippocampus activation when remembering common objects and scenes. The study team will examine differences between participants with Opioid Use Disorder (OUD) and those without OUD.
Differences in Hippocampal (Hpc) volume | Day 2 (MRI task visit)
  T-1 weighted structural images for each participant will be used to compute the volume of the hippocampus in people with OUD compared to those without OUD.
Differences in hippocampal circuit connectivity | Day 2 (MRI task visit)
  Functional connectivity, measured with BOLD signal will be used to examine functional connectivity between the hippocampus, amygdala, and prefrontal cortex. The study team will examine differences in connectivity between participants with OUD and those without OUD.
Differences in performance | Day 1 (computer tasks visit)
  Number of correct responses will be used to assess memory for common objects and scenes. Differences in memory will be examined in between participants with OUD and those without OUD.
Differences in performance | Day 2 (MRI task visit)
  Number of correct responses will be used to assess memory for common objects and scenes. Differences in memory will be examined in between participants with OUD and those without OUD.
Differences in threat reactivity measured via skin conductance response (SCR) | Day 1 (computer tasks visit)
  Electrodermal activity collected with a bioamplifier will be used to quantify physiological reactivity to threat. Event related SCR will be measured as a baseline corrected response (peak minus baseline) to cues that predict threat compared to cues that do not predict threat. Differences in SCR between participants with OUD and participants without OUD will be examined.
Differences in threat reactivity measured via skin conductance response (SCR) | Day 2 (MRI task visit)
  Electrodermal activity collected with a bioamplifier will be used to quantify physiological reactivity to threat. Event related SCR will be measured as a baseline corrected response (peak minus baseline) to cues that predicted threat on the previous day compared to cues that did not predict threat. Differences in SCR between participants with OUD and participants without OUD will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Duval, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
It is NIH policy that the results and accomplishments of the activities that it funds should be made available to the public. The principal investigator (PI) will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented, as appropriate.
Supporting Information: Study Protocol, ICF
Time Frame: When the study is completed, access to study data will be provided by the PI as requested.